CLINICAL TRIAL: NCT00659451
Title: Effects Of Losartan On Myocardial Structure And Function And On Epicardial Fat Deposition In Diabetic Hypertensive Patients With Left Ventricular: Qualitative And Quantitative Alteration
Brief Title: Effects Of Losartan On Myocardial Structure In Diabetic Hypertensive Patients With Left Ventricular
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Responsible Party: Paola Preti/MD, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNIPV002DIM2008
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Essential Hypertension; Diabetes Mellitus
Keywords: Hypertension; Diabetes mellitus; Heart
MeSH Terms: conditions — Essential Hypertension; Diabetes Mellitus; Hypertension | interventions — Losartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Experimental): Losartan
  Interventions: Drug: Losartan
- 1 (Active Comparator): Amlodipine
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Losartan — tablets; 50, 100 mg; od; 12 months
  Arms: 2
Drug: Amlodipine — tablets; 5, 10 mg; od; 12 months
  Arms: 1

SUMMARY:
The anthypertensive treatment with Losartan may have benefits beyond blood pressure reduction on myocardial structure and function in hypertensive diabetic patients. We will evaluate the effect of losartan treatment on structural characteristics of myocardium in hypertensive diabetic patients:

1. left ventricular mass, intraventricular septal thickness, fractional shortening.
2. myocardial qualitative alteration and heterogeneity of myocardial tissue that describes myocardial texture and echodensity, related to collagen deposition; myocardial qualitative alteration will be evaluate by ultrasonic myocardial integrated backscatter signals (IBS) both as peak end diastolic signal intensity and as cardiac cyclic variation
3. alteration of diastolic function as studied by Doppler flow velocities across the mitral valve (Pulse Wave Doppler) and pulse wave Tissue Doppler Imaging parameters
4. aortic strain and distensibility (that is in relation with LVH)
5. epicardial adipose tissue measurement (this parameter is related to the visceral fat and may be an easy method to indicate patients with high cardiovascular risk).

ELIGIBILITY:
Inclusion Criteria:

* Gender: 50% Male and 50 % female
* Age: 40-80 years
* Race: caucasian
* Well controlled type II Diabetes : fasting glicemia < 126 mg/dl in two different determinantion or any non fasting glicemia > 200 mg/dl; HbA1c < 7%
* Mild to moderate hypertension (BP>130/80mmHg; <160/100mmHg)
* Left ventricular hypertrophy (LVMI > 131/110 g/m2 in males/females respectively)

Exclusion Criteria:

* other anthypertensive treatment after wash out period of 2 weeks
* abnormal heart rest function (EF < 55%).
* valvular heart disease
* congenital heart disease
* heart failure or prior myocardial infarction
* renal disease
* liver disease
* connective tissue disease
* pregnancy or lactation
* sensitivity to the study drugs
* contraindication from an approved label

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mass, intraventricular septal thickness, fractional shortening; myocardial qualitative and diastolic function alteration; aortic strain and distensibility. | Between 08.00 and 10.00 at baseline, and after 3, 6, and 12 months

SECONDARY OUTCOMES:
Heterogeneity of myocardial tissue; epicardial adipose tissue measurement | Between 08.00 and 10.00 at baseline, and after 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pavia, Pavia, Italy